CLINICAL TRIAL: NCT00857012
Title: Arimidex: Compliance and Arthralgias in Clinical Therapy (COMPACT): An in Practice Assessment of Arthralgias and Related Costs as Well as Compliance in the First Year of Anastrozole Therapy
Brief Title: Arimidex: Compliance and Arthralgias in Clinical Therapy (COMPACT)
Acronym: COMPACT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ODE-ARI-2008/1
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer
Keywords: Primary early MCa; Arimidex
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: treated with Anastrozole as per SPC

SUMMARY:
Patients are eligible for inclusion in this NIS if they have taken anastrozole either upfront or following two to three years of tamoxifen treatment ("switch") for at least three and not more than six months prior to offering an individual participation in this program. Treatment should follow local therapy guidelines and standard practice. Treatment decisions for patients participating in this study including assessments or supportive therapy during follow-up visits will also follow guidelines and remain independent of the program.

DETAILED DESCRIPTION:
The patient population will include postmenopausal women with hormone-receptor positive primary breast cancer scheduled for adjuvant upfront endocrine treatment with anastrozole or following two to three years of tamoxifen treatment ("switch") according to the current SmPC (Appendix C). Patients will have taken anastrozole for at least three months and not more than six months before the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 18 years or older; Postmenopause is defined as Natural menopause with menses >1 year ago or Serum FSH (> 20 IU/ l), and E2 levels in the postmenopausal range or patients who had bilateral oophorectomy
* Histologically / cytologically confirmed primary diagnosis of early breast cancer (M0) with hormone sensitive tumour (ER+ve and/or PgR+ve)
* Patients, who underwent breast cancer surgery and, if appl. radiation therapy and/or neo/adjuvant chemotherapy and have taken adjuvant endocrine treatment with anastrozole (upfront or following two to three years of tamoxifen) min 3 max 6 months
* In case of a previous therapy with tamoxifen (switch-therapy), duration of tamoxifen treatment for at least two and up to three years.

Exclusion Criteria:

* Patients with severe renal function disorders (Creatinine clearance < 20 ml/min or Patients with moderate or severe disorders of hepatic function
* Concomitant treatment with drugs known to affect sex hormonal status and tamoxifen
* Patients with ductal carcinoma in situ (DCIS) without primary diagnosis of early breast cancer (M0)
* Evidence of any significant clinical disorder or laboratory finding which in the opinion of the investigator, makes it undesirable for the patient to participate in the program

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will include postmenopausal women with hormone-receptor positive primary breast cancer receiving adjuvant endocrine treatment with anastrozole upfront or following two to three years of tamoxifen therapy ("switch") according to the current SmPC (Appendix C). Patients will have received anastrozole treatment for at least 3 months and up to 6 months before the start of the study.
Sampling Method: Probability Sample
Enrollment: 2313 (Actual)
Dates: Start 2009-04; Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Assessment of arthralgia scores and patients' compliance within the first year of anastrozole treatment, stratified by upfront and switch therapy as well as assessment of the relationship between compliance and arthralgia scores. | 12 months

SECONDARY OUTCOMES:
Incidence of arthralgia and arthralgia characteristics within the 1st year of anastrozole therapy stratified by upfront and switch therapy and assessment of the relationship of arthralgia incidence and arthralgia characteristics to patients compliance. | 12 months
Retrospective assessment of incidence of pre-existing arthralgias before start of anastrozole treatment, stratified by upfront and switch therapy. | 12 months
Descriptive assessment of arthralgia therapy and of costs of arthralgia therapy, stratified by upfront and switch therapy. | 12 months
Identification of factors influencing and correlating to treatment-emergent arthralgias | 12 months
Assessment of safety and tolerability of anastrozole. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: H Brasch, Study Director — AstraZeneca, Germany
Locations (383):
- Germany (383):
  - Research Site, Aachen, Germany
  - Research Site, Aalen, Germany
  - Research Site, Ahaus, Germany
  - Research Site, Albstadt, Germany
  - Research Site, Altötting, Germany
  - Research Site, Alzey, Germany
  - Research Site, Amberg, Germany
  - Research Site, Apolda, Germany
  - Research Site, Aschaffenburg, Germany
  - Research Site, Aschersleben, Germany
  - Research Site, Augsburg, Germany
  - Research Site, Aurich, Germany
  - Research Site, Babenhausen, Germany
  - Research Site, Bad Dürkheim, Germany
  - Research Site, Bad Herrenalb, Germany
  - Research Site, Bad Nauheim, Germany
  - Research Site, Bad Neuenahr-Ahrweiler, Germany
  - Research Site, Bad Oeynhausen, Germany
  - Research Site, Bad Oldesloe, Germany
  - Research Site, Bad Reichenhall, Germany
  - Research Site, Bad Saarow, Germany
  - Research Site, Bad Segeberg, Germany
  - Research Site, Bad Tölz, Germany
  - Research Site, Bad Urach, Germany
  - Research Site, Bad Wildbad, Germany
  - Research Site, Bad Wildungen, Germany
  - Research Site, Bad Windsheim, Germany
  - Research Site, Baden-Baden, Germany
  - Research Site, Bamberg, Germany
  - Research Site, Bautzen, Germany
  - Research Site, Bayreuth, Germany
  - Research Site, Berlin, Germany
  - Research Site, Bexbach, Germany
  - Research Site, Biberach, Germany
  - Research Site, Biedenkopf, Germany
  - Research Site, Bielefeld, Germany
  - Research Site, Bietigheim-Bissingen, Germany
  - Research Site, Blankenburg, Germany
  - Research Site, Blumberg in Baden, Germany
  - Research Site, Bocholt, Germany
  - Research Site, Bochum, Germany
  - Research Site, Bonn, Germany
  - Research Site, Borna, Germany
  - Research Site, Bottrop, Germany
  - Research Site, Böblingen, Germany
  - Research Site, Brackenheim, Germany
  - Research Site, Bramsche, Germany
  - Research Site, Brandenburg, Germany
  - Research Site, Braunschweig, Germany
  - Research Site, Bretten, Germany
  - Research Site, Bruchsal, Germany
  - Research Site, Brühl, Germany
  - Research Site, Burg, Germany
  - Research Site, Burghausen, Germany
  - Research Site, Bühl, Germany
  - Research Site, Bünde, Germany
  - Research Site, Celle, Germany
  - Research Site, Chemnitz, Germany
  - Research Site, Cloppenburg, Germany
  - Research Site, Coburg, Germany
  - Research Site, Coesfeld, Germany
  - Research Site, Cologne, Germany
  - Research Site, Dachau, Germany
  - Research Site, Damme, Germany
  - Research Site, Datteln, Germany
  - Research Site, Demmin, Germany
  - Research Site, Dessau, Germany
  - Research Site, Dießen, Germany
  - Research Site, Dillenburg, Germany
  - Research Site, Dillingen, Germany
  - Research Site, Dinkelsbühl, Germany
  - Research Site, Ditzingen, Germany
  - Research Site, Doberlug-Kirchhain, Germany
  - Research Site, Dornstadt, Germany
  - Research Site, Dorsten, Germany
  - Research Site, Dortmund, Germany
  - Research Site, Dreieich, Germany
  - Research Site, Dresden, Germany
  - Research Site, Duisburg, Germany
  - Research Site, Düren, Germany
  - Research Site, Düsseldorf, Germany
  - Research Site, Ebermannstadt, Germany
  - Research Site, Ebersbach, Germany
  - Research Site, Eggenfelden, Germany
  - Research Site, Eisenach, Germany
  - Research Site, Ellwangen, Germany
  - Research Site, Elmshorn, Germany
  - Research Site, Emmendingen, Germany
  - Research Site, Erding, Germany
  - Research Site, Erfurt, Germany
  - Research Site, Ergolding, Germany
  - Research Site, Erkelenz, Germany
  - Research Site, Eschweiler, Germany
  - Research Site, Esens, Germany
  - Research Site, Essen, Germany
  - Research Site, Ettlingen, Germany
  - Research Site, Euskirchen, Germany
  - Research Site, Eutin, Germany
  - Research Site, Feuchtwangen, Germany
  - Research Site, Flensburg, Germany
  - Research Site, Frankenberg, Germany
  - Research Site, Frankenthal, Germany
  - Research Site, Frankfurt (Oder), Germany
  - Research Site, Frechen, Germany
  - Research Site, Freiburg im Breisgau, Germany
  - Research Site, Freising, Germany
  - Research Site, Freital, Germany
  - Research Site, Freyung, Germany
  - Research Site, Friedrichshafen, Germany
  - Research Site, Fulda, Germany
  - Research Site, Fürstenfeldbruck, Germany
  - Research Site, Fürstenwalde, Germany
  - Research Site, Fürth, Germany
  - Research Site, Garbsen, Germany
  - Research Site, Geesthacht, Germany
  - Research Site, Geilenkirchen, Germany
  - Research Site, Gelsenkirchen, Germany
  - Research Site, Georgsmarienhütte, Germany
  - Research Site, Gera, Germany
  - Research Site, Geretsried, Germany
  - Research Site, Gerlingen, Germany
  - Research Site, Gersthofen, Germany
  - Research Site, Giesen, Germany
  - Research Site, Gifhorn, Germany
  - Research Site, Gladbeck, Germany
  - Research Site, Goslar, Germany
  - Research Site, Göppingen, Germany
  - Research Site, Göttingen, Germany
  - Research Site, Gräfelfing, Germany
  - Research Site, Griesheim, Germany
  - Research Site, Gummersbach, Germany
  - Research Site, Günzburg, Germany
  - Research Site, Güstrow, Germany
  - Research Site, Haiger, Germany
  - Research Site, Halberstadt, Germany
  - Research Site, Halle, Germany
  - Research Site, Hamburg, Germany
  - Research Site, Hamelin, Germany
  - Research Site, Hamm, Germany
  - Research Site, Hanover, Germany
  - Research Site, Hartha, Germany
  - Research Site, Heide, Germany
  - Research Site, Heidelberg, Germany
  - Research Site, Heidenheim, Germany
  - Research Site, Heilbronn, Germany
  - Research Site, Heinsberg, Germany
  - Research Site, Hemmingen, Germany
  - Research Site, Henstedt-Ulzburg, Germany
  - Research Site, Heppenheim an der Bergstrasse, Germany
  - Research Site, Herborn, Germany
  - Research Site, Herbrechtingen, Germany
  - Research Site, Herdecke, Germany
  - Research Site, Herford, Germany
  - Research Site, Hermsdorf, Germany
  - Research Site, Herne, Germany
  - Research Site, Herzberg, Germany
  - Research Site, Herzberg am Harz, Germany
  - Research Site, Hessisch Oldendorf, Germany
  - Research Site, Hilchenbach, Germany
  - Research Site, Hildesheim, Germany
  - Research Site, Hillesheim, Germany
  - Research Site, Hochstadt, Germany
  - Research Site, Hof, Germany
  - Research Site, Hofheim, Germany
  - Research Site, Holzminden, Germany
  - Research Site, Homburg/Saar, Germany
  - Research Site, Hückelhoven, Germany
  - Research Site, Ilsede, Germany
  - Research Site, Ingolstadt, Germany
  - Research Site, Isny, Germany
  - Research Site, Itzehoe, Germany
  - Research Site, Jena, Germany
  - Research Site, Kahla, Germany
  - Research Site, Kalkar, Germany
  - Research Site, Karlsbad, Germany
  - Research Site, Karlsruhe, Germany
  - Research Site, Kassel, Germany
  - Research Site, Kaufbeuren, Germany
  - Research Site, Kempten, Germany
  - Research Site, Kerpen, Germany
  - Research Site, Kiel, Germany
  - Research Site, Koblenz, Germany
  - Research Site, Konstanz, Germany
  - Research Site, Korntal, Germany
  - Research Site, Königs Wusterhausen, Germany
  - Research Site, Krefeld, Germany
  - Research Site, Kreuzberg, Germany
  - Research Site, Kreuztal, Germany
  - Research Site, Krumbach, Germany
  - Research Site, Kusel, Germany
  - Research Site, Künzelsau, Germany
  - Research Site, Laatzen, Germany
  - Research Site, Lahnstein, Germany
  - Research Site, Landau, Germany
  - Research Site, Landshut, Germany
  - Research Site, Langen, Germany
  - Research Site, Langenhagen, Germany
  - Research Site, Lauf, Germany
  - Research Site, Lehrte, Germany
  - Research Site, Leichlingen, Germany
  - Research Site, Leipzig, Germany
  - Research Site, Leisnig, Germany
  - Research Site, Leonberg, Germany
  - Research Site, Leverkusen, Germany
  - Research Site, Lich, Germany
  - Research Site, Limburg, Germany
  - Research Site, Lingen, Germany
  - Research Site, Lohsa OT Weisskollm, Germany
  - Research Site, Löbau, Germany
  - Research Site, Ludwigsfelde, Germany
  - Research Site, Ludwigshafen, Germany
  - Research Site, Lübeck, Germany
  - Research Site, Lüneburg, Germany
  - Research Site, Lünen, Germany
  - Research Site, Magdeburg, Germany
  - Research Site, Mannheim, Germany
  - Research Site, Marburg, Germany
  - Research Site, Marienheide, Germany
  - Research Site, Markranstädt, Germany
  - Research Site, Marktredwitz, Germany
  - Research Site, Marl, Germany
  - Research Site, Mayen, Germany
  - Research Site, Meiningen, Germany
  - Research Site, Meissen, Germany
  - Research Site, Memmingen, Germany
  - Research Site, Mendig, Germany
  - Research Site, Mettingen, Germany
  - Research Site, Metzingen, Germany
  - Research Site, Minden, Germany
  - Research Site, Mittweida, Germany
  - Research Site, Moers, Germany
  - Research Site, Mönchengladbach, Germany
  - Research Site, Mulheim A. D. Ruhr, Germany
  - Research Site, Mutlangen, Germany
  - Research Site, Mühldorf, Germany
  - Research Site, Mühlhausen, Germany
  - Research Site, Mühlheim, Germany
  - Research Site, München, Germany
  - Research Site, Münster, Germany
  - Research Site, Nauen, Germany
  - Research Site, Naunhof, Germany
  - Research Site, Neckarsulm, Germany
  - Research Site, Netphen, Germany
  - Research Site, Neubrandenburg, Germany
  - Research Site, Neuhaus am Rennweg, Germany
  - Research Site, Neumarkt, Germany
  - Research Site, Neumünster, Germany
  - Research Site, Neuruppin, Germany
  - Research Site, Neustadt, Germany
  - Research Site, Neustadt an der Weinstraße, Germany
  - Research Site, Nienburg, Germany
  - Research Site, Nordhausen, Germany
  - Research Site, Nordhorn, Germany
  - Research Site, Nuremberg, Germany
  - Research Site, Nümbrecht, Germany
  - Research Site, Nürtingen, Germany
  - Research Site, Oberhausen, Germany
  - Research Site, Oberstdorf, Germany
  - Research Site, Ochsenfurt, Germany
  - Research Site, Offenbach, Germany
  - Research Site, Offenburg, Germany
  - Research Site, Oranienburg, Germany
  - Research Site, Osnabrück, Germany
  - Research Site, Paderborn, Germany
  - Research Site, Parchim, Germany
  - Research Site, Passau, Germany
  - Research Site, Peine, Germany
  - Research Site, Penzberg, Germany
  - Research Site, Pfinztal, Germany
  - Research Site, Pforzheim, Germany
  - Research Site, Pfullingen, Germany
  - Research Site, Pinneberg, Germany
  - Research Site, Pirmasens, Germany
  - Research Site, Plauen-Kauschwitz, Germany
  - Research Site, Pocking, Germany
  - Research Site, Potsdam, Germany
  - Research Site, Quickborn, Germany
  - Research Site, Rahden, Germany
  - Research Site, Rangsdorf, Germany
  - Research Site, Ravensburg, Germany
  - Research Site, Recklinghausen, Germany
  - Research Site, Regensburg, Germany
  - Research Site, Reinbek, Germany
  - Research Site, Remchingen, Germany
  - Research Site, Remscheid, Germany
  - Research Site, Rendsburg, Germany
  - Research Site, Reutlingen, Germany
  - Research Site, Rheine, Germany
  - Research Site, Rheinfelden, Germany
  - Research Site, Riebnitz-Damgarten, Germany
  - Research Site, Riesa, Germany
  - Research Site, Rodewisch, Germany
  - Research Site, Rodgau, Germany
  - Research Site, Rosenheim, Germany
  - Research Site, Rotenburg (Wümme), Germany
  - Research Site, Rottenburg, Germany
  - Research Site, Rottweil, Germany
  - Research Site, Rösrath, Germany
  - Research Site, Saarbrücken, Germany
  - Research Site, Saarlouis, Germany
  - Research Site, Saint Wendel, Germany
  - Research Site, Salzgitter, Germany
  - Research Site, Salzwedel, Germany
  - Research Site, Sandhausen, Germany
  - Research Site, Sayda, Germany
  - Research Site, Schalksmühle, Germany
  - Research Site, Scheibenberg, Germany
  - Research Site, Schkeuditz, Germany
  - Research Site, Schleswig, Germany
  - Research Site, Schorndorf, Germany
  - Research Site, Schönaich, Germany
  - Research Site, Schönebeck, Germany
  - Research Site, Schwabach, Germany
  - Research Site, Schwandorf in Bayern, Germany
  - Research Site, Schwäbisch Hall, Germany
  - Research Site, Schweinfurt, Germany
  - Research Site, Schwerin, Germany
  - Research Site, Schwerte, Germany
  - Research Site, Schwetzingen, Germany
  - Research Site, Sebnitz, Germany
  - Research Site, Senden, Germany
  - Research Site, Siegen, Germany
  - Research Site, Simmern, Germany
  - Research Site, Singen (Hohentwiel), Germany
  - Research Site, Solingen, Germany
  - Research Site, Sögel, Germany
  - Research Site, Sömmerda, Germany
  - Research Site, Spremberg, Germany
  - Research Site, Sprockhövel, Germany
  - Research Site, Starnberg, Germany
  - Research Site, Steglitz, Germany
  - Research Site, Stendal, Germany
  - Research Site, Stockelsdorf, Germany
  - Research Site, Stralsund, Germany
  - Research Site, Stuhr, Germany
  - Research Site, Stuttgart, Germany
  - Research Site, Sulzbach-Rosenberg, Germany
  - Research Site, Teltow, Germany
  - Research Site, Tettnang, Germany
  - Research Site, Torgau, Germany
  - Research Site, Tornesch, Germany
  - Research Site, Tübingen, Germany
  - Research Site, Uelzen, Germany
  - Research Site, Uetze, Germany
  - Research Site, Ulm, Germany
  - Research Site, Vechta, Germany
  - Research Site, Vechta-Langforden, Germany
  - Research Site, Veitshöchheim, Germany
  - Research Site, Viersen, Germany
  - Research Site, Villingen-Schwenningen, Germany
  - Research Site, Vilsbiburg, Germany
  - Research Site, Vlotho, Germany
  - Research Site, Vöhringen, Germany
  - Research Site, Völklingen, Germany
  - Research Site, Waldmünchen, Germany
  - Research Site, Walsrode, Germany
  - Research Site, Wangen, Germany
  - Research Site, Warburg, Germany
  - Research Site, Warendorf, Germany
  - Research Site, Warin, Germany
  - Research Site, Wasserburg, Germany
  - Research Site, Weiden in Der Oberpfalz, Germany
  - Research Site, Weingarten, Germany
  - Research Site, Wermelskirchen, Germany
  - Research Site, Werneck, Germany
  - Research Site, Wertheim am Main, Germany
  - Research Site, Wetzlar, Germany
  - Research Site, Wiesbaden, Germany
  - Research Site, Wilster, Germany
  - Research Site, Wismar, Germany
  - Research Site, Witten, Germany
  - Research Site, Witterda, Germany
  - Research Site, Wolfen, Germany
  - Research Site, Wolfsburg, Germany
  - Research Site, Worms, Germany
  - Research Site, Wuppertal, Germany
  - Research Site, Würselen, Germany
  - Research Site, Würzburg, Germany
  - Research Site, Zittau, Germany
  - Research Site, Zossen, Germany
  - Research Site, Zwickau, Germany
  - Research Site, Zwiesel, Germany
  - Research Site, Zwönitz, Germany

REFERENCES:
- [Derived] Hadji P, Jackisch C, Bolten W, Blettner M, Hindenburg HJ, Klein P, Konig K, Kreienberg R, Rief W, Wallwiener D, Zaun S, Harbeck N. COMPliance and Arthralgia in Clinical Therapy: the COMPACT trial, assessing the incidence of arthralgia, and compliance within the first year of adjuvant anastrozole therapy. Ann Oncol. 2014 Feb;25(2):372-7. doi: 10.1093/annonc/mdt513. Epub 2013 Dec 18. PMID 24355487